CLINICAL TRIAL: NCT00160927
Title: Microcirculation cutanée et Vasodilatation Induite Par la Pression Non-Nociceptive Chez Les diabètiques
Brief Title: Microvascular Response in Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Alfediam (Other); UNIVALOIRE (Unknown)
Other Study IDs: PHRC 02-03
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2007-03-19 (Estimated); Status verified 2007-03

CONDITIONS: Diabetes Mellitus
Keywords: microcirculation; Laser doppler flowmetry; neuropathy; endothelial function
MeSH Terms: conditions — Diabetes Mellitus | interventions — Iontophoresis; Nitroprusside

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: local heating
Device: iontophoresis
Drug: actylcholine
Drug: sodium nitroprusside

SUMMARY:
Vascular and neurological mechanisms are both likely to be involved in foot ulcer. We recently reported on the hand an original transient pressure-induced vasodilation (PIV) during a 5 mmHg/min increase of pressure strain using laser Doppler flowmetry. This physiological response to non noxious external local pressure strain is a widely protective cutaneous mechanism. The impairment of PIV in diabetic subjects may be relevant to the high prevalence of foot ulcer that occurs in these individuals. The aim of the project is to analyse the different physiopathological processes involved in PIV impairment in diabetic subjects as compared to matched controls.

DETAILED DESCRIPTION:
The whole study is a prospective observational study of diabetic type 1 and type 2 subjects focusing on the various physical, physiopathological or pharmacological mechanisms that may interfere with the normal response of the cutaneous microcirculation.The study is currently conducted under various parallel groups of patients and control subjects matched on age and sexe. Techniques used for the study are only non-invasive investigations such as iontophoresis with laser doppler flowmetry, clinical and paraclinical non-invasive investigation of peripheral neuropathy, ultrasound imaging of peripheral arteries.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes

Exclusion Criteria:

* Non diabetic neuropathy
* Peripheral arterial disease
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2003-01; Study Completion 2008-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis Saumet, MD PhD, Principal Investigator — Centre Hospitalier Universitaire Angers
Locations (1):
- Centre hospitalier universitaire, Angers, France

REFERENCES:
- [Background] Koitka A, Legrand-Fernandez MS, Abraham P, Fizanne L, Fromy B, Sigaudo-Roussel D, Saumet JL. Low skin temperature impairs the cutaneous vasodilator response to local progressive pressure strain. Microvasc Res. 2004 Mar;67(2):203-6. doi: 10.1016/j.mvr.2003.12.001. PMID 15020212
- [Background] Koitka A, Abraham P, Bouhanick B, Sigaudo-Roussel D, Demiot C, Saumet JL. Impaired pressure-induced vasodilation at the foot in young adults with type 1 diabetes. Diabetes. 2004 Mar;53(3):721-5. doi: 10.2337/diabetes.53.3.721. PMID 14988257